CLINICAL TRIAL: NCT05203510
Title: A Phase 4, Prospective, Multicenter, Single-Arm Study of a Mean Pulmonary Artery Pressure-Targeted Approach With Early and Rapid Treprostinil Therapy to Reverse Right Ventricular Remodeling in Patients With Pulmonary Arterial Hypertension: ARTISAN (Afterload Reduction To Improve Right Ventricular Structure And FuNction)
Brief Title: A Study of a Mean Pulmonary Artery Pressure-Targeted Approach With Early and Rapid Treprostinil Therapy to Reverse Right Ventricular Remodeling in Participants With Pulmonary Arterial Hypertension
Acronym: ARTISAN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Collaborators: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REM-PH-418
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treprostinil (Experimental): Participants will receive parenteral treprostinil at initial dose of 1.25 nanograms/kilogram/minute (at minimum) either intravenously or subcutaneously. Based on mPAP assessments and after a minimum dose of parenteral treprostinil is reached, at Investigator's (PI's) discretion, participants may transition to oral treprostinil and continue dose uptitration for further reduction of mPAP. Based on Month 12 mPAP assessment, participants may transition from parenteral to oral treprostinil at PI's discretion after completion of Month 12 assessment and continue uptitration for further reduction of mPAP. If minimum dose of parenteral treprostinil is not reached at Month 6/12 at PI's discretion, uptitration of parenteral treprostinil or oral treprostinil transition may occur to maintain normal mPAP.
  Treprostinil therapy (parenteral or oral) may continue as tolerated toward goal of further reduction of mPAP until Month 36.
  Interventions: Drug: Parenteral Treprostinil; Drug: Oral Treprostinil

INTERVENTIONS:
Drug: Parenteral Treprostinil — Parenteral treprostinil will be administered per schedule specified in the arm description.
  Other Names: Remodulin
Drug: Oral Treprostinil — Oral treprostinil will be administered per schedule specified in the arm description.
  Other Names: Orenitram

SUMMARY:
The primary objective of this study is to assess the effect of early and rapid treprostinil therapy for mean pulmonary artery pressure (mPAP) reduction to improve right ventricular (RV) function and reverse RV remodeling in participants with pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PAH (WHO Group 1) classified by one of the following subgroups:

  * Idiopathic, heritable or drug/toxin induced (with the exception of amphetamine-induced PAH)
  * Associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥1 year)
  * Associated with connective tissue disease
  * Associated with human immunodeficiency virus infection
* Baseline visit right heart catheterization (RHC) must also meet the following criteria:

  * mPAP >35 mmHg
  * Pulmonary vascular resistance (PVR) >2 Wood units
  * Pulmonary artery wedge pressure (PAWP) ≤15 mmHg
* On a stable dose of an endothelin receptor antagonist (ERA) and/or phosphodiesterase type 5 inhibitor (PDE-5i) or soluble guanylate cyclase stimulator (sGC) therapy or if treatment naïve, willing to take one of these medications in addition to study drug
* REVEAL Lite 2 risk score ≤9
* WHO FC II or III
* 6MWD >165 meters

Exclusion Criteria:

PAH-related Exclusion Criteria:

* Prior or current use of epoprostenol, treprostinil, iloprost, beraprost, or selexipag
* Positive vasoreactivity test in idiopathic, heritable, or drug/toxin induced PAH
* Amphetamine use within the past 12 months
* WHO Groups 2, 3, 4, and 5
* Use of any other investigational drug, device, or therapy within 30 days of the Baseline visit
* Moderate or severe hepatic impairment (Child-Pugh Class B and C)
* Any other clinically significant illness or abnormal laboratory value(s) measured during screening that, in the opinion of the Investigator, might adversely affect interpretation of the study data or participant safety (for example, active infection, chronic thromboembolic pulmonary hypertension, or acute/recent deep vein thrombosis or pulmonary embolism)
* Chronic atrial fibrillation, multiple premature ventricular or atrial contractions of clinical significance, or any other condition that would interfere with proper cardiac gating during cMRI
* Permanent cardiac pacemaker or automatic internal cardioverter that would interfere with conduct of cMRI
* Metallic implant (for example, defibrillator, neurostimulator, hearing aid, permanent infusion device, implantable pump, or body plates/screws/bolts) that would interfere with conduct of cMRI

CardioMEMS-related Exclusion Criteria, if applicable:

* Previously implanted with CardioMEMS pulmonary artery Sensor or unwilling/unable to permit collection and perform upload (transmission) of pulmonary artery pressure (PAP) readings
* Unable to take dual antiplatelet or anticoagulation therapy for 30 days after CardioMEMS PA Sensor implantation unless the participant has an indication for warfarin or direct oral anticoagulant

NOTE: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Right Ventricular Ejection Fraction (RVEF), as Measured by Cardiac Magnetic Resonance Imaging (cMRI) at Month 12 | Baseline, Month 12

SECONDARY OUTCOMES:
Change From Baseline in mPAP at Month 12 | Baseline, Month 12
Number of Participants With Clinical Improvement From Baseline to Month 12, 24, and 36 | Baseline to Months 12, 24, and 36
  Clinical improvement is defined as meeting all 3 criteria: - improvement in six-minute walk distance (6MWD) increase ≥10% or ≥30 meters; - improvement in World Health Organization (WHO) functional class (FC) or maintenance of WHO FC I/II; - improvement in N-terminal pro-brain natriuretic peptide (NT-proBNP) decrease ≥30% or <300 ng/liter (L).
Change From Baseline in RV-Pulmonary Artery (PA) Coupling Estimated by the Ratio of Stroke Volume by End Systolic Volume at Month 12 | Baseline, Month 12
Change From Baseline in RV End-Diastolic Volume Index at Month 12 | Baseline, Month 12
Change From Baseline in RV Stroke Volume Index at Month 12 | Baseline, Month 12
Change From Baseline in 6MWD at Month 12, 24, and 36 | Baseline, Months 12, 24, and 36
Change From Baseline in Registry to EValuate EArly and Long-Term PAH Disease Management (REVEAL) Lite 2 Risk Score at Months 12, 24, and 36 | Baseline, Months 12, 24, and 36
Change From Baseline in WHO FC at Months 12, 24, and 36 | Baseline, Months 12, 24, and 36
Change From Baseline in NT-proBNP at Months 12, 24, and 36 | Baseline, Months 12, 24, and 36
Change From Baseline in Borg Dyspnea Score at Months 12, 24, and 36 | Baseline, Months 12, 24, and 36
Change From Baseline in RV-PA Coupling Estimated by the Ratio of Tricuspid Annular Plane Systolic Excursion by Pulmonary Artery Systolic Pressure (TAPSE/PASP) at Months 12, 24, and 36 | Baseline, Months 12, 24, and 36
Survival Rate: Number of Participants who Survived at Months 12, 24, and 36 | Baseline to Months 12, 24, and 36
Change From Baseline in mPAP at Months 24 and 36 | Baseline, Months 24 and 36

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Banner University Medical Center (University of Arizona), Phoenix, Arizona
  - HonorHealth John C. Lincoln Medical Center, Phoenix, Arizona
  - University of California San Francisco - Fresno, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco Pulmonary, Critical Care, Allergy and Sleep Medicine, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - USF, Tampa, Florida
  - Georgia Clinical Research, Austell, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Health North Hospital, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Temple Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Carilion Clinic, Roanoke, Virginia